CLINICAL TRIAL: NCT03661996
Title: An Open-label, 8-Week Study to Compare the Comfort and Ease of Use of Five Different Treatment Regimens for CNTX-4975-05 Intra-articular Injection in Subjects With Chronic, Moderate-to-Severe Osteoarthritis Knee Pain
Brief Title: An Open-label, 8-week Safety, Efficacy, and Assessment of Cooling Methods for Administration of CNTX-4975-05 for Knee OA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centrexion Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CNTX-4975i-OA-303
Record Dates: First submitted 2018-08-28; First posted 2018-09-07 (Actual); Results first posted 2022-03-09 (Actual); Last update posted 2022-03-09 (Actual); Status verified 2022-01

CONDITIONS: Knee Osteoarthritis
Keywords: osteoarthritis; knee pain; non opioid; analgesic; capsaicin; pain; intra-articular
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis; Pain | interventions — Capsaicin; Lidocaine; Epinephrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Breg Cooling Control Group (Experimental): Subject receives 2% lidocaine and CNTX-4975-05 with cooling device Breg ice water pump.
  Interventions: Drug: CNTX-4975-05; Drug: Lidocaine without epinephrine; Device: Breg Ice Water Pump
- Gel Pack Cooling Group (Experimental): Subject receives 2% lidocaine and CNTX-4975-05 with cooling device Elasto-Gel.
  Interventions: Drug: CNTX-4975-05; Drug: Lidocaine without epinephrine; Device: ElastoGel
- Shortened Gel Pack Cooling Group (Experimental): Subject receives 2% lidocaine and CNTX-4975-05 with cooling device Elasto-Gel.
  Interventions: Drug: CNTX-4975-05; Drug: Lidocaine without epinephrine; Device: ElastoGel
- Single Needle Injection Gel Pack Cooling Group - 2% Lidocaine (Experimental): Subject receives 2% lidocaine and CNTX-4975-05 with cooling device Elasto-Gel.
  Interventions: Drug: CNTX-4975-05; Drug: Lidocaine without epinephrine; Device: ElastoGel
- Single Needle Injection Gel Pack Cooling Group - 1% Lidocaine (Experimental): Subject receives 1% lidocaine and CNTX-4975-05 with cooling device Elasto-Gel.
  Interventions: Drug: CNTX-4975-05; Drug: Lidocaine without epinephrine; Device: ElastoGel

INTERVENTIONS:
Drug: CNTX-4975-05 — Osteoarthritis (OA) intra-articular injection of CNTX-4975-05
  Other Names: capsaicin
Drug: Lidocaine without epinephrine — 15 mL lidocaine intra-articular injection
  Other Names: Lidocaine
Device: ElastoGel — Cooling Device
  Arms: Gel Pack Cooling Group; Shortened Gel Pack Cooling Group; Single Needle Injection Gel Pack Cooling Group - 1% Lidocaine; Single Needle Injection Gel Pack Cooling Group - 2% Lidocaine
Device: Breg Ice Water Pump — Cooling Device
  Arms: Breg Cooling Control Group

SUMMARY:
An Open-label, 8-Week Study to Compare the Comfort and Ease of Use of Five Different Treatment Regimens for CNTX 4975-05 Intra-articular Injection in Subjects with Chronic, Moderate-to-Severe Osteoarthritis Knee Pain.

DETAILED DESCRIPTION:
This is an open-label, single injection (per knee), 8-week study to evaluate the comfort and ease of use of 5 different treatment regimens, and to evaluate the efficacy and safety of a single intra-articular (IA) injection, in one or both knees, of CNTX-4975-05 in subjects with chronic, moderate-to-severe knee OA pain. Procedural pain associated with IA injection of the investigational product, CNTX-4975-05, will be controlled primarily through adjunct controlled joint cooling and secondarily by pre-medication with IA lidocaine.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or female subjects between 40 and 95 years of age (inclusive)
* Confirmation of osteoarthritis (OA) of the knee: radiography of both knees using standard standing films (scored by the investigator) or using the fixed flexion method, taken during the Screening Visit of CNTX-4975i-OA-301 or CNTX-4975i-OA-304.
* Confirmation of OA of the index knee: American College of Rheumatology (ACR) diagnostic criteria
* For subjects for monoarticular knee injection, the index knee must have moderate to severe pain at screening associated with OA, which must be stable for a minimum of 6 months prior to Screening, as assessed by the investigator.

These subjects may have:

1. unilateral or bilateral OA, with the index knee having moderate to severe pain, and the contralateral knee having none to mild pain, OR
2. unilateral or bilateral OA, with the index knee having moderate to severe pain and the other knee having had a PJR or TJR within 5 years of the Screening Visit. The knee with the PJR/TJR is not to be injected with CNTX-4975-05.

For subjects for bilateral knee injection, the index knee must have moderate to severe pain at screening associated with OA, and greater pain in the index knee than in the contralateral knee. Their pain must be stable for a minimum of 6 months prior to Screening, as assessed by the investigator. The index knee in these subjects is the one with the worst pain with walking. Where both knees have equal pain with walking, then the knee on the subject's dominant side will be designated the index knee.

For qualifying knee pain with walking, subjects will use an NPRS (0-10; 0=no pain, 10=worst possible pain) to rate their knee pain with walking (both knees, except knees with PJR/TJR). The PJR/TJR pain should be rated using the NPRS scale, but will not be a qualifying pain score.

* Body mass index ≤45 kg/m^2.

Key Exclusion Criteria:

* Joint replacement surgery of the index knee at any time, or open surgery of the index knee in the past 24 months. Joint replacement of the contralateral knee is permitted for subjects who will not receive an injection in the contralateral (natural) knee.
* Prior arthroscopic surgery of the index knee within 6 months of Screening.
* Any painful conditions of the index knee due to joint disease other than OA. Radicular or referred pain involving the index knee or from joint disease other than OA involving the index knee, such as, but not restricted to chondromalacia patellae, inflammatory disease, metabolic diseases, gout/pseudogout, hemochromatosis, acromegaly, etc.
* Periarticular pain from any cause, including referred pain, bursitis, tendonitis, soft tissue tenderness, or subacute/acute pain from injury.
* Other chronic pain anywhere in the body that requires the use of chronic analgesic medications, including, but not limited to, local painful areas, myofascial pain syndromes, fibromyalgia, genetic, metabolic abnormalities, hematologic, or neuropathic pain.

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 854 (Actual)
Dates: Start 2018-09-18 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Randall M. Stevens, MD, Study Chair — Centrexion Therapeutics Corp
Locations (28):
- United States (28):
  - Alabama Orthopaedic Center-Research, Birmingham, Alabama
  - Holland Center for Family Health, Peoria, Arizona
  - Noble Clinical Research, Tucson, Arizona
  - Med Center Medical Clinic, Carmichael, California
  - Core Healthcare Group, Cerritos, California
  - Encompass Clinical Research, Spring Valley, California
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Conquest Clinical Research, Maitland, Florida
  - F&T Medical Research, Inc., Miami, Florida
  - M&M Medical Center, Inc., Miami, Florida
  - Charter Research, Mt. Dora, Florida
  - Premier MED Family & Sports Medicine, Ocoee, Florida
  - Ascension Research, Pinellas Park, Florida
  - M&M Clinical Trials Sunrise, Sunrise, Florida
  - Georgia Institute for Clinical Research, LLC, Marietta, Georgia
  - Atlanta Orthopaedic Institute, LLC, Stockbridge, Georgia
  - Healthcare Research Network II, LLC, Flossmoor, Illinois
  - Affinity Health, Oak Brook, Illinois
  - MediSphere Medical Research Center, LLC, Evansville, Indiana
  - Tandem Clinical Research, Marrero, Louisiana
  - DelRicht Research, New Orleans, Louisiana
  - Healthcare Research Network, Hazelwood, Missouri
  - Center for Pharmaceutical Research, LLC, Kansas City, Missouri
  - Office of Robert P. Kaplan, DO, Las Vegas, Nevada
  - Hassman Research Institute, Berlin, New Jersey
  - First Surgical Hospital, Bellaire, Texas
  - Metroplex Clinical Research Center, Dallas, Texas
  - Hermann Drive Surgical Hospital, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited between 18 September 2018 and 22 October 2019
Groups:
- Group 1. Breg Cooling Control: Breg Cooler (total cool time at least 85 minutes) with IA injection of 2% lidocaine followed by a second IA injection CNTX-4975
- Group 2. Gel Pack Cooling: Gel Pack Cooling (total cool time at least 60 minutes) with IA injection of 2% lidocaine followed by a second IA injection CNTX-4975
- Group 3. Shortened Gel Pack Cooling: Gel pack cooling (total cool time at least 35 minutes) with IA injection of 2% lidocaine followed by a second IA injection CNTX-4975
- Group 4. Single Needle Injection Gel Pack Cooling - 2% Lidocaine: Gel pack cooling (total cool time at least 45 minutes) with a combined single IA injection of 2% lidocaine followed by CNTX-4975
- Group 5. Single Needle Injection Gel Pack Cooling - 1% Lidocaine: Gel pack cooling (total cool time at least 45 minutes) with a combined single IA injection of 1% lidocaine followed by CNTX-4975
Period: Overall Study
Arm/Group | Group 1. Breg Cooling Control | Group 2. Gel Pack Cooling | Group 3. Shortened Gel Pack Cooling | Group 4. Single Needle Injection Gel Pack Cooling - 2% Lidocaine | Group 5. Single Needle Injection Gel Pack Cooling - 1% Lidocaine
Started | 162 | 180 | 176 | 163 | 173
Treated | 162 | 179 | 175 | 160 | 172
Completed | 150 | 172 | 170 | 150 | 159
Not Completed | 12 | 8 | 6 | 13 | 14
Not completed — Adverse Event | 0 | 0 | 1 | 1 | 0
Not completed — Lost to Follow-up | 5 | 1 | 2 | 2 | 6
Not completed — Physician Decision | 1 | 1 | 1 | 2 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 3 | 5 | 1 | 7 | 7
Not completed — Sponsors Decision | 2 | 0 | 0 | 0 | 0
Not completed — Other | 1 | 1 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Population, all subjects who received any amount of CNTX-4975-05
Groups:
- Group 1. Breg Cooling Control: The subject received intra-articular injections from separate needles of 2% lidocaine without epinephrine followed by CNTX-4975-05 15 minutes later. The subject was cooled with the Breg ice water pump and circumferential knee wrap for 15 minutes before lidocaine injection, followed by 30 minutes before the CNTX-4975-05 injection, and for at least 30 minutes and up to 90 minutes after the CNTX-4975-05 injection as needed.
- Group 2. Gel Pack Cooling: The subject received intra-articular injections from separate needles of 2% lidocaine without epinephrine followed by CNTX-4975-05 10 minutes later. The subject was cooled with the Elasto-Gel circumferential knee wrap for 40 minutes before the lidocaine injection, followed by 10 minutes before the CNTX-4975-05 injection, and for at least 10 minutes and up to 90 minutes after the CNTX-4975-05 injection as needed.
- Group 3. Shortened Gel Pack Cooling: The subject received intra-articular injections from separate needles of 2% lidocaine without epinephrine followed by CNTX-4975-05 5 minutes later. The subject was cooled with the Elasto-Gel circumferential knee wrap for 30 minutes before the lidocaine injection, followed by 5 minutes before the CNTX-4975-05 injection, and with no required cooling after the CNTX-4975-05 injection, but up to 90 minutes of cooling as needed.
- Group 4. Single Needle Injection Gel Pack Cooling - 2% Lidocaine: The subject received intra-articular injections from a single needle of 2% lidocaine without epinephrine and CNTX-4975-05, with up to 3 minutes in between injections. The subject was cooled with the Elasto-Gel circumferential knee wrap for 45 minutes before the single needle injection of lidocaine and CNTX-4975-05. There was no cooling in between injections and no cooling required after the single needle injections, but up to 90 minutes of cooling as needed.
- Group 5. Single Needle Injection Gel Pack Cooling - 1% Lidocaine: The subject received intra-articular injections from a single needle of 1% lidocaine without epinephrine and CNTX-4975-05, with up to 3 minutes in between injections. The subject was cooled with the Elasto-Gel circumferential knee wrap for 45 minutes before the single needle injection of lidocaine and CNTX-4975-05. There was no cooling in between injections and no cooling required after the single needle injections, but up to 90 minutes of cooling as needed.
- Total: Total of all reporting groups
Arm/Group | Group 1. Breg Cooling Control | Group 2. Gel Pack Cooling | Group 3. Shortened Gel Pack Cooling | Group 4. Single Needle Injection Gel Pack Cooling - 2% Lidocaine | Group 5. Single Needle Injection Gel Pack Cooling - 1% Lidocaine | Total
Number analyzed (Participants) | 162 | 179 | 175 | 160 | 172 | 848
Age, Continuous [Mean (Standard Deviation); unit: Years] | 62.2 (9.5) | 61.8 (8.8) | 63.9 (9.2) | 62.6 (9.4) | 65.1 (9.9) | 63.1 (9.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 104 | 101 | 104 | 99 | 100 | 508
  Male | 58 | 78 | 71 | 61 | 72 | 340
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 69 | 88 | 15 | 17 | 7 | 196
  Not Hispanic or Latino | 93 | 91 | 160 | 143 | 164 | 651
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Body Mass Index (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] | 31.21 (5.349) | 29.94 (5.276) | 31.89 (7.904) | 31.54 (6.083) | 31.72 (6.099) | 31.25 (6.252)
Radiographic Osteoarthritis Type [Count of Participants; unit: Participants]
  Unilateral | 9 | 43 | 31 | 22 | 50 | 155
  Bilateral | 153 | 136 | 144 | 138 | 122 | 693
Subject Type [Count of Participants; unit: Participants]
  Single Knee Injection (Unilateral Mod-Sec OA Knee Pain) | 26 | 50 | 71 | 57 | 69 | 273
  Single knee Injection (Non-Index knee PJR/TJR) | 3 | 12 | 12 | 9 | 16 | 52
  Bilateral Knee Injections (Bilateral mod-Sec OA Knee Pain) | 133 | 117 | 92 | 94 | 87 | 523
KOOS Pain Subscale (Index Knee) [Mean (Standard Deviation); unit: score on a scale] — The KOOS (KOOS = Knee Injury and Osteoarthritis Outcome Score) was developed as an extension of the WOMAC (Western Ontario and McMaster Universities Arthritis Index) to evaluate the dimensions of knee osteoarthritis associated pain and injury. It includes 5 separately scored subscales: Pain, Symptoms (including stiffness), Function (Daily Living), Function (Sports and Recreational Activities), and knee-related Quality of Life. Each subscale score is rated on a 5-point scale (i.e., 0 to 4). Higher scores indicate better outcome.
  score on a scale | 42.42 (12.959) | 44.89 (13.397) | 48.30 (15.071) | 44.70 (12.803) | 44.33 (14.201) | 44.97 (13.830)
KOOS Symptoms Subscale (Index Knee) [Mean (Standard Deviation); unit: score on a scale] — The KOOS (KOOS = Knee Injury and Osteoarthritis Outcome Score) was developed as an extension of the WOMAC (Western Ontario and McMaster Universities Arthritis Index) to evaluate the dimensions of knee osteoarthritis associated pain and injury. It includes 5 separately scored subscales: Pain, Symptoms (including stiffness), Function (Daily Living), Function (Sports and Recreational Activities), and knee-related Quality of Life. Each subscale score is rated on a 5-point scale (i.e., 0 to 4). Higher scores indicate better outcome.
  score on a scale | 47.69 (16.611) | 50.86 (16.161) | 52.75 (17.570) | 47.97 (14.484) | 51.73 (16.227) | 50.26 (16.348)
KOOS Function (Daily Living) Subscale (Index Knee) [Mean (Standard Deviation); unit: score on a scale] — The KOOS (KOOS = Knee Injury and Osteoarthritis Outcome Score) was developed as an extension of the WOMAC (Western Ontario and McMaster Universities Arthritis Index) to evaluate the dimensions of knee osteoarthritis associated pain and injury. It includes 5 separately scored subscales: Pain, Symptoms (including stiffness), Function (Daily Living), Function (Sports and Recreational Activities), and knee-related Quality of Life. Each subscale score is rated on a 5-point scale (i.e., 0 to 4). Higher scores indicate better outcome.
  score on a scale | 46.42 (13.586) | 47.81 (13.791) | 52.50 (15.846) | 48.87 (14.535) | 47.05 (14.511) | 48.55 (14.607)
KOOS Function (Sport and Recreational Activities) Subscale (Index Knee) [Mean (Standard Deviation); unit: score on a scale] — The KOOS (KOOS = Knee Injury and Osteoarthritis Outcome Score) was developed as an extension of the WOMAC (Western Ontario and McMaster Universities Arthritis Index) to evaluate the dimensions of knee osteoarthritis associated pain and injury. It includes 5 separately scored subscales: Pain, Symptoms (including stiffness), Function (Daily Living), Function (Sports and Recreational Activities), and knee-related Quality of Life. Each subscale score is rated on a 5-point scale (i.e., 0 to 4). Higher scores indicate better outcome.
  score on a scale | 25.06 (18.485) | 23.44 (19.417) | 26.29 (21.980) | 30.66 (23.312) | 30.74 (24.279) | 27.12 (21.747)
KOOS Quality of Life Subscale (Index Knee) [Mean (Standard Deviation); unit: score on a scale] — The KOOS (KOOS = Knee Injury and Osteoarthritis Outcome Score) was developed as an extension of the WOMAC (Western Ontario and McMaster Universities Arthritis Index) to evaluate the dimensions of knee osteoarthritis associated pain and injury. It includes 5 separately scored subscales: Pain, Symptoms (including stiffness), Function (Daily Living), Function (Sports and Recreational Activities), and knee-related Quality of Life. Each subscale score is rated on a 5-point scale (i.e., 0 to 4). Higher scores indicate better outcome.
  score on a scale | 31.98 (16.387) | 36.31 (17.450) | 30.24 (16.751) | 32.93 (18.248) | 27.54 (16.620) | 31.83 (17.313)
Pain with Walking NPRS (0-10) Score [Mean (Standard Deviation); unit: score on a scale] — The pain with walking Numerical Pain Rating Scale (NPRS) (0-10, 0 being no pain, 10 being greatest pain) collected subjects' average pain with walking over the past 24 hours. Subjects recorded the pain in their target knee, either the index knee or additionally the non-index knee in the case of bilateral subjects.
  Lower scores indicate less pain, higher scores indicate higher pain.
  score on a scale | 7.58 (1.413) | 7.23 (1.311) | 6.70 (1.585) | 6.83 (1.493) | 6.91 (1.367) | 7.05 (1.467)

OUTCOME MEASURES:

1. Primary Outcome: Determination of Optimal Procedure for Administering CNTX-4975-05 With Regards to Pain, Participant Satisfaction, and Investigator's Satisfaction
Description: A composite score was calculated for each of the 5 treatment regimens by summing the scores of three assessments: (1) procedure pain 30 minutes after injection of CNTX-4975-05 on a 0-4 scale, 0 was best indicating no procedure pain, 4 was worst indicating severe procedure pain; (2) assessment of subjects' satisfaction with the regimen on a scale of 1 (completely dissatisfied) to 7 (completely satisfied), 1 was worst and 7 was best; and (3) assessment of investigators' satisfaction with the regimen on a scale of 1 (completely dissatisfied) to 7 (completely satisfied), 1 was worst and 7 was best.
  The procedure pain at 30 minutes was reversed to a 1-7 scale so 7 was best indicating no procedure pain and 1 was worst indicating severe procedure pain. The three assessments were summed for a total score from 3-21, 3 being the worst outcome and 21 being the best outcome. The geometric mean of the scores was derived for each group.
  All assessments were administered on Day 1 (Baseline).
Time Frame: Day 1 assessments
Population: The intent to treat (ITT) population included all enrolled subjects who received any amount of CNTX-4975-05. A subject was considered enrolled if they had a Treatment Day 1 study visit.
Measure: Geometric Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Group 1. Breg Cooling Control | Group 2. Gel Pack Cooling | Group 3. Shortened Gel Pack Cooling | Group 4. Single Needle Injection Gel Pack Cooling - 2% Lidocaine | Group 5. Single Needle Injection Gel Pack Cooling - 1% Lidocaine
Number analyzed (Participants) | 162 | 179 | 175 | 160 | 172
score on a scale | 17.18 (1.016) | 18.26 (1.015) | 16.48 (1.016) | 17.40 (1.016) | 16.00 (1.015)
Statistical Analysis 1: Comparison: Group 1. Breg Cooling Control vs Group 2. Gel Pack Cooling; Geometric LS means, ratio of geometric LS means, with Breg Cooling as control, and 95% CIs were obtained from an ANCOVA model on the natural log-transformed composite outcome with cooling and injection procedure as the main effect. Baseline K-L grade, baseline BMI category, sex, and reverse-scored and normalized index knee procedure pain were included as covariates. Estimates and CIs on the log scale were exponentiated to obtain ratios of geometric means on the original scale; Test type: Non-Inferiority — The treatment regimen is Clinically Acceptable if it is no more than 30% worse than the Breg Cooling Control Group and the lower bound of the 95% CI for Ratio of Geometric LS Means is greater than 0.7; Ratio of Geometric LS Means = 1.063, 95% CI 2-sided [1.019 to 1.108], Standard Error of Mean 1.0216 — Parameter dispersion is the Standard Error of the Ratio of Geometric LS Means
Statistical Analysis 2: Comparison: Group 1. Breg Cooling Control vs Group 3. Shortened Gel Pack Cooling; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Ratio of Geometric LS Means = 0.959, 95% CI 2-sided [0.919 to 1.001], Standard Error of Mean 1.0221 — Parameter dispersion is the Standard Error of the Ratio of Geometric LS Means
Statistical Analysis 3: Comparison: Group 1. Breg Cooling Control vs Group 4. Single Needle Injection Gel Pack Cooling - 2% Lidocaine; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Ratio of Geometric LS Means = 1.013, 95% CI 2-sided [0.970 to 1.057], Standard Error of Mean 1.0219 — Parameter dispersion is the Standard Error of the Ratio of Geometric LS Means
Statistical Analysis 4: Comparison: Group 1. Breg Cooling Control vs Group 5. Single Needle Injection Gel Pack Cooling - 1% Lidocaine; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority — [test comment as in outcome 1, analysis 1]; Ratio of Geometric LS Means = 0.931, 95% CI 2-sided [0.892 to 0.972], Standard Error of Mean 1.0219 — Parameter dispersion is the Standard Error of the Ratio of Geometric LS Means

2. Secondary Outcome: Mean Change From Baseline in KOOS "Symptoms" Subscale Score by Subject Type
Description: The KOOS (KOOS = Knee Injury and Osteoarthritis Outcome Score) was developed as an extension of the WOMAC (Western Ontario and McMaster Universities Arthritis Index) to evaluate the dimensions of knee osteoarthritis associated pain and injury. It includes 5 separately scored subscales: Pain, Symptoms (including stiffness), Function (Daily Living), Function (Sports and Recreational Activities), and knee-related Quality of Life. Each subscale score is rated on a 5-point scale (i.e., 0 to 4). The previous week is the time period evaluated when answering the questions. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
  The KOOS was administered on Day 1 (Baseline) and Week 8.
  Higher scores (or positive change from baseline) indicate improvement.
Time Frame: Baseline, Week 8
Population: The intent to treat (ITT) population included all enrolled subjects who received any amount of CNTX-4975-05.A subject was considered enrolled if they had a Treatment Day 1 study visit.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE: Subjects with moderate to severe OA knee pain in the index knee and mild to no pain in the non-index knee; results reported for the index knee
- Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE: Subjects with single knee OA pain in the index knee and a partial or total knee joint replacement in the non-index knee; results reported for index knee
- Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE: Subjects with moderate to severe knee OA pain in both the index and non-index knee; results reported for the index knee in these subjects
- Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE: Subjects with moderate to severe knee OA pain in both the index and non-index knee that received bilateral injections of CNTX-4975; results reported for the non-index knee in these subjects
Arm/Group | Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE | Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE
Number analyzed (Participants) | 260 | 50 | 492 | 381
score on a scale | 17.15 (1.396) | 20.41 (3.692) | 20.05 (0.981) | 18.40 (1.011)
Statistical Analysis 1: Comparison: Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE; Results are summarized by subject type and the injected knee. The KOOS subscale scores are derived and normalized. Higher scores indicate improvement. Model terms included pooled site group, baseline K-L grade category, baseline BMI category, sex, study visit, and baseline subscale score as covariates; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 17.15, 95% CI 2-sided [14.40 to 19.90], Standard Error of Mean 1.396
Statistical Analysis 2: Comparison: Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Mean Difference (Final Values) = 20.41, 95% CI 2-sided [12.79 to 28.03], Standard Error of Mean 3.692
Statistical Analysis 3: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 20.05, 95% CI 2-sided [18.44 to 21.66], Standard Error of Mean 0.819
Statistical Analysis 4: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 18.40, 95% CI 2-sided [16.41 to 20.38], Standard Error of Mean 1.011

3. Secondary Outcome: Mean Change From Baseline in KOOS "Pain" Subscale Score by Subject Type
Description: as for outcome 2
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE | Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE
Number analyzed (Participants) | 260 | 50 | 488 | 379
score on a scale | 22.45 (1.478) | 23.90 (4.613) | 25.62 (0.865) | 22.10 (1.053)
Statistical Analysis 1: Comparison: Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 22.45, 95% CI 2-sided [19.54 to 25.37], Standard Error of Mean 1.478
Statistical Analysis 2: Comparison: Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 23.90, 95% CI 2-sided [14.38 to 33.42], Standard Error of Mean 4.613
Statistical Analysis 3: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 25.62, 95% CI 2-sided [23.92 to 27.32], Standard Error of Mean 0.865
Statistical Analysis 4: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 22.10, 95% CI 2-sided [20.03 to 24.17], Standard Error of Mean 1.053

4. Secondary Outcome: Mean Change From Baseline in KOOS "Pain With Walking" Single Question Score by Subject Type
Description: The KOOS (KOOS = Knee Injury and Osteoarthritis Outcome Score) was developed as an extension of the WOMAC (Western Ontario and McMaster Universities Arthritis Index) to evaluate the dimensions of knee osteoarthritis associated pain and injury. It includes 5 separately scored subscales: Pain, Symptoms (including stiffness), Function (Daily Living), Function (Sports and Recreational Activities), and knee-related Quality of Life. Each subscale score is rated on a 5-point scale (i.e., 0 to 4). The previous week is the time period evaluated when answering the questions. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. The KOOS Pain with Walking is a single question from the KOOS Pain subscale.
  The KOOS was administered on Day 1 (Baseline) and Week 8.
  Higher scores (or positive change from baseline) indicate improvement.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE | Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE
Number analyzed (Participants) | 260 | 50 | 488 | 379
score on a scale | 21.08 (1.744) | 25.26 (6.062) | 25.85 (1.035) | 23.34 (1.238)
Statistical Analysis 1: Comparison: Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE; Results are summarized by subject type and the injected knee. The KOOS subscale scores are derived and normalized. Higher scores indicate improvement. Model terms for pooled site group, baseline K-L grade category, baseline BMI category (<30 kg/m2, ≥30 kg/m2), sex, study visit, and baseline KOOS subscale score as covariates. Study visit was included in the model as a categorical variable; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 21.1, 95% CI 2-sided [17.6 to 24.5], Standard Error of Mean 1.74
Statistical Analysis 2: Comparison: Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p = 0.0003, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 25.3, 95% CI 2-sided [12.7 to 37.8], Standard Error of Mean 6.06
Statistical Analysis 3: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 25.85, 95% CI 2-sided [23.82 to 27.88], Standard Error of Mean 1.035
Statistical Analysis 4: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE; [analysis description as in outcome 4, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 23.34, 95% CI 2-sided [20.91 to 25.78], Standard Error of Mean 1.238

5. Secondary Outcome: Mean Change From Baseline in KOOS "Function (Daily Living)" Subscale Score by Subject Type
Description: The KOOS (KOOS = Knee Injury and Osteoarthritis Outcome Score) was developed as an extension of the WOMAC (Western Ontario and McMaster Universities Arthritis Index) to evaluate the dimensions of knee osteoarthritis associated pain and injury. It includes 5 separately scored subscales: Pain, Symptoms (including stiffness), Function (Daily Living), Function (Sports and Recreational Activities), and knee-related QOL. Each subscale score is rated on a 5-point scale (i.e., 0 to 4). The previous week is the time period evaluated when answering the questions. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale.
  The KOOS was administered on Day 1 (Baseline) and Week 8.
  Higher scores (or positive change from baseline) indicate improvement.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE | Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE
Number analyzed (Participants) | 260 | 50 | 487 | 379
score on a scale | 20.86 (1.481) | 25.66 (4.568) | 25.57 (0.861) | 22.26 (1.058)
Statistical Analysis 1: Comparison: Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 20.86, 95% CI 2-sided [17.94 to 23.78], Standard Error of Mean 1.481
Statistical Analysis 2: Comparison: Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 25.66, 95% CI 2-sided [16.24 to 35.09], Standard Error of Mean 4.568
Statistical Analysis 3: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 25.57, 95% CI 2-sided [23.88 to 27.26], Standard Error of Mean 0.861
Statistical Analysis 4: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 25.69, 95% CI 2-sided [24.02 to 27.37], Standard Error of Mean 0.853

6. Secondary Outcome: Mean Change From Baseline in KOOS "Function (Sport and Recreational Activities)" Subscale Score by Subject Type
Description: as for outcome 5
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE | Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE
Number analyzed (Participants) | 255 | 49 | 482 | 375
score on a scale | 25.17 (2.248) | 33.11 (5.795) | 27.80 (1.233) | 24.80 (1.598)
Statistical Analysis 1: Comparison: Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 25.17, 95% CI 2-sided [20.74 to 29.60], Standard Error of Mean 2.248
Statistical Analysis 2: Comparison: Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 33.11, 95% CI 2-sided [21.15 to 45.07], Standard Error of Mean 5.795
Statistical Analysis 3: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 27.80, 95% CI 2-sided [25.38 to 30.23], Standard Error of Mean 1.233
Statistical Analysis 4: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 24.80, 95% CI 2-sided [21.66 to 27.94], Standard Error of Mean 1.598

7. Secondary Outcome: Mean Change From Baseline in KOOS "Knee-Related Quality of Life" Subscale Score by Subject Type
Description: as for outcome 5
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE | Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE
Number analyzed (Participants) | 260 | 50 | 488 | 379
score on a scale | 22.10 (1.898) | 16.75 (6.255) | 21.52 (1.062) | 19.40 (1.365)
Statistical Analysis 1: Comparison: Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 22.10, 95% CI 2-sided [18.37 to 25.84], Standard Error of Mean 1.898
Statistical Analysis 2: Comparison: Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 16.75, 95% CI 2-sided [3.84 to 29.66], Standard Error of Mean 6.255
Statistical Analysis 3: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 21.52, 95% CI 2-sided [19.43 to 23.60], Standard Error of Mean 1.062
Statistical Analysis 4: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE; [analysis description as in outcome 2, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = 19.40, 95% CI 2-sided [16.72 to 22.09], Standard Error of Mean 1.365

8. Secondary Outcome: Mean Change From Baseline in Average Daily Pain With Walking NPRS (0-10) Score by Subject Type
Description: The pain with walking Numerical Pain Rating Scale (NPRS) (0-10, 0 being no pain, 10 being greatest pain) collected subjects' average pain with walking over the past 24 hours. Subjects recorded the pain in their target knee, either the index knee or additionally the non-index knee in the case of bilateral subjects. The NPRS was collected at Day 1 (Baseline) and Week 8.
  Lower scores (or negative change from baseline) indicate improvement
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE | Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE
Number analyzed (Participants) | 260 | 51 | 491 | 414
score on a scale | -3.48 (0.191) | -3.52 (0.416) | -4.02 (0.118) | -3.72 (0.122)
Statistical Analysis 1: Comparison: Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) INDEX KNEE; Results are summarized by subject type and the injected knee. The NPRS was collected during the last study visit. Lower scores indicate improvement. Model terms included pooled site group, baseline K-L grade category, baseline BMI category, sex, study visit, and baseline pain score as covariates; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = -3.48, 95% CI 2-sided [-3.86 to -3.10], Standard Error of Mean 0.191
Statistical Analysis 2: Comparison: Single Knee Injection (Non-Index Knee PJR/TJR) INDEX KNEE; [analysis description as in outcome 8, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = -3.52, 95% CI 2-sided [-4.38 to -2.67], Standard Error of Mean 0.416
Statistical Analysis 3: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) INDEX KNEE; [analysis description as in outcome 8, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = -4.02, 95% CI 2-sided [-4.25 to -3.79], Standard Error of Mean 0.118
Statistical Analysis 4: Comparison: Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) NON-INDEX KNEE; [analysis description as in outcome 8, analysis 1]; Test type: Superiority — A within-group analysis of change at Week 8 from baseline; p < 0.0001, Mixed Models Analysis; LS means, 95% CIs, and P values were obtained from a mixed model for repeated measures (MMRM); Least Squares Mean Change From Baseline = -3.72, 95% CI 2-sided [-3.96 to -3.48], Standard Error of Mean 0.122

ADVERSE EVENTS:
Time Frame: Adverse events were collected from Screening to the End of the Study (8 Weeks)
Description: Adverse events are reported here according to bilateral or unilateral injection group. Adverse events by injection group is of greater safety consequence and interest than events by cooling regimens because the injection group delineates exposures to CNTX-4975-05 (index knee only or bilateral intra-articular injections) while the cooling regimens does not. Therefore representing adverse events by injection group is a better indicator of safety in relation to study drug.
Groups:
- Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) Day 1 Through Week 8/Early Termination: Subjects with moderate to severe OA knee pain in the index knee and mild to no pain in the non-index knee; TEAEs presented for subjects in the Single Knee Injection groups represents TEAEs occurring from Day 1 through Week 8/Early Termination
- Single Knee Injection (Non-Index Knee PJR/TJR) Day 1 Through Week 8/Early Termination: Single Knee Injection (Non-index Knee partial or total joint replacement)
  Data presented for subjects in the Single Knee Injection groups represents TEAEs occurring from Day 1 through Week 8/Early Termination
- Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) Day 1 Through Day 7: Subjects with moderate to severe knee OA pain in both the index and non-index knee; TEAEs presented for subjects in the Bilateral Knee Injection group only from Day 1 (index knee) through Day 7 (i.e., prior to them receiving the second intra-articular injection of CNTX-4975)
- Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) Day 7 Through Week 8/Early Termination: Subjects with moderate to severe knee OA pain in both the index and non-index knee that received bilateral injections of CNTX-4975; TEAEs presented for subjects in the Bilateral Knee Injection group from Day 8 (i.e., after receiving the second injection of CNTX-4975 into the nonindex knee) to Week 8/Early Termination. Note: 96 subjects did not receive a second injection of CNTX-4975
Arm/Group | Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) Day 1 Through Week 8/Early Termination | Single Knee Injection (Non-Index Knee PJR/TJR) Day 1 Through Week 8/Early Termination | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) Day 1 Through Day 7 | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) Day 7 Through Week 8/Early Termination
All-Cause Mortality (participants affected / at risk) | 0/273 | 0/52 | 0/523 | 0/427
Serious Adverse Events (participants affected / at risk) | 1/273 | 0/52 | 0/523 | 5/427
Other Adverse Events (participants affected / at risk) | 33/273 | 11/52 | 18/523 | 27/427
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) Day 1 Through Week 8/Early Termination (N=273) | Single Knee Injection (Non-Index Knee PJR/TJR) Day 1 Through Week 8/Early Termination (N=52) | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) Day 1 Through Day 7 (N=523) | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) Day 7 Through Week 8/Early Termination (N=427)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Atrial Fibrillation (Cardiac disorders) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 0 | 0 | 1
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 0.1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Knee Injection (Unilateral Mod-Sev OA Knee Pain) Day 1 Through Week 8/Early Termination (N=273) | Single Knee Injection (Non-Index Knee PJR/TJR) Day 1 Through Week 8/Early Termination (N=52) | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) Day 1 Through Day 7 (N=523) | Bilateral Knee Injection (Bilateral Mod-Sev OA Knee Pain) Day 7 Through Week 8/Early Termination (N=427)
Back Pain (Musculoskeletal and connective tissue disorders) | 5 | 2 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 1 | 0 | 3
Joint Swelling (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2 | 2
Muscle Spasm (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 2
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 3 | 0
Abdominal Upper Pain (Gastrointestinal disorders) | 2 | 0 | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 0
Nasopharyngitis (Infections and infestations) | 2 | 0 | 2 | 5
Bronchitis (Infections and infestations) | 1 | 1 | 0 | 0
Upper Respiratory tract infectiosn (Infections and infestations) | 1 | 1 | 0 | 0
Cellulitis (Infections and infestations) | 0 | 0 | 0 | 2
Urinary Track Infection (Infections and infestations) | 0 | 0 | 0 | 2
Ligament Sprain (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Skin abrasion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Puritus (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0
Alanine aminotransferase (Investigations) | 2 | 0 | 0 | 0
Blood creatine increased (Investigations) | 0 | 0 | 0 | 2
Headache (Nervous system disorders) | 1 | 1 | 2 | 3
Tooth extraction (Vascular disorders) | 1 | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 2
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-06-13): https://cdn.clinicaltrials.gov/large-docs/96/NCT03661996/Prot_SAP_000.pdf